CLINICAL TRIAL: NCT02970448
Title: Expedited Laser Interstitial Thermal Therapy and Chemoradiation for Patients With Newly Diagnosed High Grade Gliomas
Brief Title: Expedited Laser Interstitial Thermal Therapy + Chemoradiation For Newly Diagnosed High Grade Gliomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4316
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: High Grade Glioma
Keywords: LITT; Brain Tumor; Temozolomide
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- LITT with Radiation and Temozolomide (Experimental): Laser interstitial thermal therapy (LITT) followed by Radiation therapy, three-dimensional conformal radiotherapy (3D-CRT) or intensity modulation radiation therapy (IMRT), 60 Gy/30 fractions. Radiation given with chemotherapy Temozolomide
  Interventions: Procedure: LITT; Radiation: Radiation therapy; Drug: Temozolomide

INTERVENTIONS:
Procedure: LITT — MRI-guided laser interstitial thermal therapy uses a gas cooled side-firing (directional) laser and a variety of procedure specific tools to thermally ablate target tissue in-situ.
  Other Names: Laser interstitial thermal therapy
Radiation: Radiation therapy — One treatment of 2 Gy will be given daily 5 days per week for a total of 60 Gy over 6 weeks. All portals shall be treated during each treatment session. Doses are specified such that at least 95% of the planning target volume (PTV) shall receive 100% of the prescribed dose.
  Other Names: 3D-Conformal radiation therapy (RT); Intensity Modulated RT
Drug: Temozolomide — Temozolomide will be administered continuously from day 1 of radiotherapy to the last day of radiation at a daily oral dose of 75 mg/m2 for a maximum of 49 days

SUMMARY:
The investigators of this study want to see if shortening the total treatment time for brain tumors is safe.The treatment for participant's brain tumors is laser surgery (Laser Interstitial Thermal Therapy (LITT)) followed by radiation with chemotherapy. For participants, the total time of treatment from surgery to the end of radiation and chemotherapy is about l 0 weeks long. This study asks whether it is safe to shorten the total treatment to 7 weeks.

To shorten the total treatment time, investigators want to see if it is safe to start radiation with chemotherapy within 5 days after surgery. Usually patients start their radiation with chemotherapy about 21-28 days after the surgery.

Shortening the total time of treatment may allow investigators to kill the cancer cells more effectively.

DETAILED DESCRIPTION:
Primary Objective To determine the safety and feasibility of reducing the time interval between LITT and the start of chemoradiation to ≤ 7 days.

The primary endpoint (binary) for safety/feasibility will be defined as the occurrence of one or more of the following within each patient during a window of observation from the completion LITT to the end of radiation:

* Wound dehiscence, grade 3 {CTCAE v4.0)
* Seizures, grade 3 (CTCAE v4.0) in patients without a prior history of seizures and on adequate anti-seizure medications
* Cerebral edema, grade 4 (CTCAE v4.0)
* Failure to complete of 60 Grays (Gy) of radiation

Secondary Objective(s) To estimate the proportion of patients requiring adjustments in radiation plans post-LITT.

Secondary Endpoint: Requirement of an adjustment in the radiation plan to account for post-LITT tissue distortion.

Study design This study will be a 2-stage, single-institution safety and feasibility trial. Patients will be evaluated by a neuro-oncology team consisting of a neurosurgeon trained in LITT, radiation oncologist and medical oncologist prior to surgery. Evaluable patients will have a histologic diagnosis of high-grade glioma, complete LITT, and are candidates for standard concurrent radiation (60 Gy) and temozolomide as determined by the treating physician. Concurrent chemoradiation will begin within 7 days of the LITT procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have suspected high grade glioma by MRI
* Subjects must have received no prior therapies for this disease.
* Patients must be considered appropriate candidates for LITT.
* Karnofsky Performance status ≥ 60%
* Subjects must have normal organ and marrow function as defined below. Measures of function must be within 14 days prior to registration.

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3, platelets ≥ 100,000 cells/mm3, hemoglobin ≥ 10.0 g/dl. Use of transfusion or other intervention to achieve this hemoglobin level is acceptable.
  * Blood urea nitrogen ≤ 30mg/dl and creatinine ≤ 1.7 mg/dl
  * Bilirubin ≤ 2.0 mg/dl, Aspartate aminotransferase/ Alanine aminotransferase (AST/ALT) ≤ 3x upper limit of normal
  * Electrocardiogram without evidence of acute cardiac ischemia
  * Prothrombin time/international normalized ratio (PT INR) <1.4
* Women of childbearing potential and male participants must practice adequate contraception.
* For women of childbearing age, negative pregnancy test within 14 days prior to registration
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants not eligible to obtain MRI with and without contrast
* Recurrent High grade gliomas (HGG)
* Cerebral edema, grade 3 or greater prior to surgery
* Post-operative complications including significant neurological decline or hemorrhage that causes a drop in KPS to less than 60 or renders the patient not suitable for chemoradiation as determined by their treating physician
* Severe co-morbidity that would confer excess risk of surgery, radiation or chemotherapy, as determined by the treating physician.

Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration of completion of protocol therapy

* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Participants receiving other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Study safety as determined by the number of patients who experience pre-specified adverse events | Up to 12 weeks after LITT therapy
  pre-specified adverse events include: Wound dehiscence, grade 3 (CTCAE v4.0), Grade 3 Seizures (CTCAE v4.0) in patients without a prior history of seizures and on adequate anti-seizure medications, Cerebral edema, grade 4 (CTCAE v4.0), Failure to complete of 60 Gy radiation

SECONDARY OUTCOMES:
Number of patients with adjustments to radiation plan to account for post-LITT tissue distortion | Up to 12 weeks after LITT therapy
  The proportion of patients requiring a change in radiation plan after fusion of the plan with the post-operative MRI will be calculated, and a 95% confidence interval will be placed on this proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Yu, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States